CLINICAL TRIAL: NCT03736733
Title: Relevance of an Adapted and Supervised Physical Activity Program in Fibromyalgia Patients. The FIMOUV 1 Study. Interventional, Controlled, Randomized, Open Study of an Original Outpatient Management.
Brief Title: Relevance of an Adapted and Supervised Physical Activity Program in Fibromyalgia Patients. The FIMOUV 1 Study.
Acronym: FIMOUV 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18CH051; 2018-A01597-48 (Other: ANSM)
Record Dates: First submitted 2018-11-05; First posted 2018-11-09 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-02

CONDITIONS: Fibromyalgia; Physical Activity
Keywords: sedentary time
MeSH Terms: conditions — Fibromyalgia; Motor Activity; Sedentary Behavior | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fibromyalgia patients with physical activity program (Experimental): Two weekly exercise sessions at the university hospital of St-Etienne for 1 month then relay outside in a sports association or club certified "Sports Health" in the Loire (42) or Haute-Loire (43) for 2 months.
  Interventions: Other: physical activity program
- fibromyalgia patients with physical activity at home (Other): Advice and recommendations of physical activity at home (= current clinical practice, from 1 to 3 sessions per week in autonomy).
  Interventions: Other: Advice and recommendations of physical activity at home

INTERVENTIONS:
Other: physical activity program — Two weekly exercise sessions at the university hospital of St-Etienne for 1 month then relay outside in a sports association or club certified "Sports Health" in the Loire (42) or Haute-Loire (43) for 2 months.
  Arms: fibromyalgia patients with physical activity program
Other: Advice and recommendations of physical activity at home — Advice and recommendations of physical activity at home (= current clinical practice, from 1 to 3 sessions per week in autonomy).
  Arms: fibromyalgia patients with physical activity at home

SUMMARY:
Fibromyalgia affects 2 to 5% of adults in the general population. Patients describe a combination of symptoms centred around fatigue not induced by exercise and not relieved by rest.

The diagnosis of fibromyalgia is self-perpetuating by the deconditioning, consequence of a reduced muscle mass due to inactivity and periods of prolonged rest.

Thus, it seems fundamental to develop other non-drug approaches: among them, adapted physical activity is recommended by most learned societies because of a good level of evidence (Level 1, Grade A). The question remains, however, whether simple advice to resume physical activity is sufficient (routine care with medical assessment at 3 months) or whether a physical activity supervised inside and outside the hospital is not more relevant.

ELIGIBILITY:
Inclusion Criteria:

* Patient lived in t Loire (42) or Haute-Loire (43)
* Patient diagnosed with fibromyalgia according to ACR (American College of rheumatology) criteria (total score WPI (Widespread Pain Index) + SS (Severity Scale) ) ≥ 13
* French writing and speaking
* Sedentary or low level of activity (less than 2 hours of regular physical activity per week at the time of inclusion)
* Signature of informed consent

Exclusion Criteria:

* Cardiac or respiratory diseases that contraindicate the practice of physical activity
* Significant co-morbidities that contraindicate the practice of physical activity: associated cardiac pathologies (severe rhythm disorders such as rapid atrial fibrillation), respiratory pathologies (severe obstructive or severe respiratory insufficiency), disabling joint pathologies (knee osteoarthritis or osteoarthritis of the hip) training on a treadmill or on a high intensity bike).
* Impossibility of submitting to the medical monitoring of the program for geographical, social or psychological reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2021-06-11 (Actual)

PRIMARY OUTCOMES:
Assessment of the impact of a 3-month program | at 3 months
  Health status assessed by the PGIC = Patient Global Impression of Change. interpretation : 0= no change, 7= clear improvement, 5= better).

SECONDARY OUTCOMES:
fatigue | at 3 months
  assessed by Fatigue Severity Scale. This is a short questionnaire of 9 questions to which the patient answers on a scale from 1 to 7.
  Simply add the scores and divide by 9 - you get a result on 7 points. The higher the result, the greater the fatigue. Several studies speak of a threshold at 5.5
Quality of sleep | at 3 months
  assessed by the Pittsburgh. The questionnaire includes 19 self-assessment questions and 5 questions for the spouse or roommate (if any). Only self-assessment questions are included in the score.
  The 19 self-assessment questions combine to give 7 components" of the score with each component receiving a score of 0 to 3.
  In all cases, a score of 0 indicates that there is no difficulty while a score of 3 indicates the existence of severe difficulties. The 7 components of the score add up to give an overall score from 0 to 21 points, 0 meaning that there is no difficulty, and 21 indicating on the contrary major difficulties.
Anxiety and Depression | at 3 months
  assessed by the Hospital Anxiety and Depression Scale (HADS) : An overall score of 19 or more indicates a major depressive episode. An overall score of 13 corresponds to adjustment disorders and minor depression.
pain catastrophizing | at 3 months
  assessed by the PCS (pain catastrophizing scale) assessing catastrophism : there are thirteen statements describing different thoughts and emotions that may be associated with pain. the person must indicate how painful these thoughts and emotions are. From 0= not at all to 4 = all the time
pain evaluation | at 3 months
  assessed by analog visual evaluation of pain (0= no pain and 10 = very painful)
muscle power | at 3 months
  evaluated by dynamometry on a stress platform (arms and legs) and by a pocket dynamometer.
muscular endurance | at 3 months
  evaluated by dynamometry on a stress platform (arms and legs).
gas exchange measurement | at 3 months
  evaluated during a stress test
quantification of physical activity in meter-h/week | at 3 months
  evaluated by the APAQ : Adult Physical Activity Questionnaire
sedentary times in hours/day | at 3 months
  evaluated by the APAQ : Adult Physical Activity Questionnaire
daily energy expenditure | at 3 months
  evaluated by actimetry
time of physical activity | at 3 months
  evaluated by actimetry
physical inactivity | at 3 months
  evaluated by actimetry
patient adherence | at 3, 6 and 12 months
  number of sessions performed
Direct medical costs | at 3, 6 and 12 months
  consultations, examinations, hospitalizations in euros
Direct non-medical costs | at 3, 6 and 12 months
  transport
Cost of lost productivity | at 3, 6 and 12 months
  time not worked

CONTACTS AND LOCATIONS:
Overall Officials: David HUPIN, MD, Principal Investigator — CHU de Saint Etienne
Locations (1):
- Chu Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No